CLINICAL TRIAL: NCT06467461
Title: Identification of Prodromal Neurodegeneration in Serotonergic-Induced REM Sleep Behavior Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NEUR-2023-32484
Record Dates: First submitted 2024-06-10; First posted 2024-06-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Dementia With Lewy Bodies; Parkinson Disease; REM Sleep Behavior Disorder
MeSH Terms: conditions — Lewy Body Disease; Parkinson Disease; REM Sleep Behavior Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research participants (Other): Adults under the age of 75; who do not meet criteria for Parkinson's disease, dementia with Lewy bodies, Alzheimer's disease, other diagnosed neurodegenerative disorder, or other known cause of RBD; and have a history of or currently use the SSRIs of interest.
  Interventions: Diagnostic Test: Skin biopsy; Diagnostic Test: Speech testing; Diagnostic Test: Ultra high field 7T MRI

INTERVENTIONS:
Diagnostic Test: Skin biopsy — Skin biopsy to detect systemic alpha-synuclein pathology in 5-HT RBD
Diagnostic Test: Speech testing — Speech Testing to quantify evolving signs of 5-HT RBD
Diagnostic Test: Ultra high field 7T MRI — 7T MRI to examine 5-HT RBD for evidence of brainstem neurodegeneration

SUMMARY:
This project will test the hypotheses that people with 5-HT RBD have systemic alpha- synuclein pathology, prodromal DLB signs, and brainstem lesions in regions that control REM sleep. AIM 1 will seek to detect abnormally phosphorylated alpha- synuclein aggregates on targeted skin biopsy in a cohort of people with 5-HT RBD and matched controls (taking SSRIs but without RBD). Aim 2 will use ultra-high field MRI at 7T to examine the pontine region of the coeruleus/subcoeruleus complex for evidence of neurodegeneration as well as segment and parcellate REM sleep related neuronal structures. Aim 3 will test for speech deficits. While these aims are independent we suspect that the severity of autonomic, speech and cognitive deficits will correlate with loss of neuromelanin signal on MRI and pathology on skin biopsy.

The investigation is a longitudinal designed study to examine histopathology, neuroimaging changes and speech function from baseline (Time 1) to a follow-up after 30 months (Time 2). A total of 60 individuals, 30 with 5-HT RBD and 30 controls, will be recruited at Time 1, brought back at Time 2, and tested across all Aims at both study visits.

ELIGIBILITY:
Inclusion Criteria:

Serotonergic REM sleep behavior (5-HT RBD) participants

Inclusion Criteria:

* Diagnosis of polysomnogram-confirmed RBD with history of dream enactment or clear dream enactment visualized on video from polysomnogram.
* History of dream enactment began shortly after (less than 2 months) starting a serotonergic antidepressant medication. Control Participants

Inclusion Criteria:

* Age (±3 years) and sex matched to participants with 5-HT RBD
* On serotonergic medication for at least 6 months without history of dream enactment.

The following serotonergic medications will be included:

Citalopram, Escitalopram, Fluoxetine, Fluvoxamine, Paroxetine, and Sertraline

Exclusion Criteria:

Serotonergic REM sleep behavior (5-HT RBD) participants

Exclusion Criteria:

* Younger than 18
* Older than 75
* Meet criteria for Parkinson's disease, dementia with Lewy bodies, Multiple System Atrophy, Pure Autonomic Failure, Alzheimer's disease, other diagnosed neurodegenerative disorder, or other known cause of RBD (e.g. narcolepsy)
* Untreated obstructive sleep apnea, obesity hypoventilation, central sleep apnea or other sleep disordered breathing
* History of dysarthria, aphasia or other condition which could interfere with speech assessment
* Reduced capacity to consent
* MRI exclusion criteria for 7T scans: presence of any metallic clip(s) or implantable medical devices (e.g., heart valve, aneurysm clip, coils or surgery, renal or aortic clips, shunts, stents or stent grafts, metal mesh/coil implants, neurostimulator, insulin pump, IVC filter, etc.).
* History of allergic response to xylocaine or other local anesthesia
* Pregnant women will be excluded due to unknown risk of MRI on developing fetus Control Participants

Exclusion Criteria: same exclusion criteria as 5-HT RBD group, plus the following:

* History of dream enactment that may suggest RBD
* Increased REM motor tone (REM atonia index > 0.10) on PSG suggestive of RBD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Phosphorylated alpha synuclein deposits on skin biopsy | time point 1 (baseline) and time point 2 (24 months, +/- 3 months)
  Incidence (positive or negative) of phosphorylated alpha synuclein deposits. Indicating direct histopathological confirmation of underlying alpha-synuclein degeneration in 5-HT RBD in a cohort of people with 5-HT RBD and matched controls (taking SSRIs but without RBD).
Neuromelanin signal intensity in the Subcoeruleus/Coeruleus Complex | time point 1 (baseline) and time point 2 (24 months, +/- 3 months)
  Examination of the pontine region of the coeruleus/subcoeruleus complex for evidence of neurodegeneration as well as segment and parcellate REM sleep related neuronal structures.
Monopitch as measured by fundamental frequency variability. | time point 1 (baseline) and time point 2 (24 months, +/- 3 months)
  Participants' voice and speech quality will be examined for synucleinopathy syndrome. The focus on speech function is designed to detect subtle brainstem deficits prior to more overt manifestations of cortical dementia.

SECONDARY OUTCOMES:
Subject-specific masks of all REM sleep-related pontine nuclei of interest, volume of Subcoeruleus/Coeruleus Complex. | time point 1 (baseline) and time point 2 (24 months, +/- 3 months)
  Subject-specific masks of all REM sleep-related pontine nuclei of interest, volume of Subcoeruleus/Coeruleus Complex.
Speed of articulatory change as measured by F2 Transitions | time point 1 (baseline) and time point 2 (24 months, +/- 3 months)
  Speed of articulatory change as measured by F2 Transitions, which are shown to be reduced in people with dysarthria

CONTACTS AND LOCATIONS:
Overall Officials: Michael Howell, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States